CLINICAL TRIAL: NCT05132309
Title: Study of Influence of Chronic Pancreatitis Severity Degree With Possible Complication of Pancreatic External Secretory Insufficiency on Intestinal Microbiota Composition Patterns
Brief Title: Intestinal Microbiota Composition in Patients With Chronic Pancreatitis and Pancreatic Exocrine Insufficiency
Status: Completed | Type: Observational
Sponsor: Federal Research and Clinical Center of Physical-Chemical Medicine (Other)
Collaborators: Moscow State University of Medicine and Dentistry (Other)
Responsible Party: Sponsor
Other Study IDs: CP-2021
Record Dates: First submitted 2021-07-30; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-08

CONDITIONS: Chronic Pancreatitis; Pancreatic Exocrine Insufficiency
MeSH Terms: conditions — Pancreatitis, Chronic; Exocrine Pancreatic Insufficiency | interventions — Enzyme Replacement Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Chronic pancreatitis without pancreatic external insufficiency
  Interventions: Combination Product: enzyme replacement therapy
- Chronic pancreatitis with mild pancreatic external insufficiency
  Interventions: Combination Product: enzyme replacement therapy
- Chronic pancreatitis with severe pancreatic external insufficiency
  Interventions: Combination Product: enzyme replacement therapy
- Chronic pancreatitis with severe pancreatic external insufficiency who underwent pancreatic surger
  Interventions: Combination Product: enzyme replacement therapy

INTERVENTIONS:
Combination Product: enzyme replacement therapy — Correction of the previously prescribed dose of enzyme replacement therapy (ERT)/first time selection of ERT according to the severity of pancreatic exocrine insufficiency

SUMMARY:
Assessment of qualitative and quantitative composition of the intestinal microbiota in patients with CP; in patients with CP and PEI complication of mild to severe degree; patients with CP and PEI who underwent surgical intervention on the pancreas. Intergroup comparison of the microbial compositional characteristics and their analysis. Correction of enzyme replacement therapy in selected groups of patients with regard to the identified microbial characteristics. Assessment of the intestinal microbiota composition in dynamics after 6 (+1) months on the background of allocated therapy

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years old; any gender;
* Chronic pancreatitis etiology: idiopathic, biliary dependent, drug-induced, alcoholic, dysmetabolic, CP as a consequence of recurrent and severe acute pancreatitis (postnecrotic);
* History of confirming diagnostic criteria of CP (in accordance with 1) Clinical guidelines of the Russian Gastroenterological Association on the diagnosis and treatment of exocrine pancreatic insufficiency 2018; 2) Clinical guidelines of the unified European guidelines for gastroenterology, on the diagnosis and therapy of chronic pancreatitis 2017; 3) Clinical guidelines of the American College of Gastroenterology 2020);
* CP diagnosis according to multispiral computed tomography of the abdominal cavity and/or endoscopic ultrasonography of pancreas: size changes; dilatation of the main pancreatic duct more than 2 mm; increased echogenicity of the walls, uneven contours and heterogeneity of the BP parenchyma, concrements or calcification of the parenchyma;
* Clinical manifestations of exocrine insufficiency of pancreas: stool disorders (mushy/liquid stool, number of defecation acts >3 p/day, undigested food remains), steatorrhea, abdominal distention, nausea/vomiting, weight loss progression with adequate caloric intake and no other objective reasons of weight loss;
* Fecal elastase-1 values less than 200 µg/g (for CP groups with EPI) or more than 200 µg/g (for CP group without concomitant EPI);
* Informed patient consent to participate in the study.

Exclusion Criteria:

* Acute pancreatitis;
* Hepatitis, cirrhosis of any etiology;
* Any acid-dependent diseases requiring immediate or long-term proton pump inhibitor therapy (PPI): gastroesophageal reflux disease, acute gastroduodenal erosions of any etiology; Zollinger-Ellison syndrome, etc;
* Stenosis of pylorys or duodenum;
* Condition after gastric resection or gastrectomy;
* Obstructive and autoimmune CP;
* Mesenteric ischemia syndrome;
* Any other cause of chronic diarrhea (irritable bowel syndrome with diarrhea predominance, gluten enteropathy, lactase deficiency, inflammatory bowel disease, etc.);
* Concomitant administration of drugs directly affecting exocrine pancreatic secretion (octreotide);
* Any concomitant diseases in the stage of decompensation (cardiovascular, renal failure, diabetes mellitus, etc.);
* Chronic infectious diseases requiring constant (long-term) supportive therapy, including HIV infection, etc;
* Hypersensitivity to pancreatin;
* Use of pro-, pre-, synbiotics, week prior to inclusion in this study;
* Use of antibiotics within 4 weeks prior to inclusion in this study;
* Pregnancy and lactation;
* Use of prohibited concomitant therapy during the study: pro-, pre-, synbiotics, including dietary fiber preparations and lactulose, as well as antibiotics, intestinal antiseptics, loperamide, intestinal sorbents.

Ages: 23 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Genetic study of fecal samples of patients with CP | 1 week
  Fecal samples of patients with CP from selected patient groups with/without PEI meet inclusion criteria will undergo 16s rRNA gene sequencing for further comparative intergroup analysis of the obtained data.
Genetic study of fecal samples of patients with CP | 6 months
  Fecal samples of patients with CP from selected patient groups with/without PEI meet inclusion criteria will undergo 16s rRNA gene sequencing for further comparative intergroup analysis of the obtained data.
Analysis of intestinal microbiota composition of patients with CP receiving 40,000 units of pancreatin per meal per day | 6 months
  Analysis of intestinal microbiota composition of patients with CP from selected patient groups with/without PEI receiving adequate dosage of enzyme replacement therapy: 40,000 units of pancreatin per meal per day
Analysis of intestinal microbiota composition of patients with CP receiving inadequate dosage of pancreatin per meal per day | 6 month
  Analysis of intestinal microbiota composition of patients with CP from selected patient groups with/without PEI receiving inadequate dosage of enzyme replacement therapy: (less then adequate dosage) of pancreatin per meal per day

CONTACTS AND LOCATIONS:
Overall Officials: Elena Ilina, Prof, Study Director — Federal Research and Clinical Center of Physical-Chemical Medicine; Igor Maev, Prof, Study Director — Moscow State University of Medicine and Dentistry
Locations (2):
- Russia (2):
  - Federal Research and Clinical Center of Physical-Chemical Medicine, Moscow (FRCC PCM), Moscow
  - Moscow State University of Medicine and Dentistry, Moscow